CLINICAL TRIAL: NCT01439490
Title: Feasibility Study: FES-PET to Determine ER-expression in Epithelial Ovarian Cancer
Brief Title: FES-PET to Determine ER-expression in Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: RUG2011-0704
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- FES-PET (Experimental): Patients undergo FES-PET prior to obtaining histology
  Interventions: Other: FES-PET

INTERVENTIONS:
Other: FES-PET — Patients undergo FES-PET prior to obtaining histology

SUMMARY:
Estrogens are implicated in the development of ovarian cancer and estrogen receptors (ER) alpha and beta are present in 20-100% of ovarian cancer patients. For this reason, antihormonal therapy with anti-estrogens or ER-antagonists is potentially an attractive treatment option. However, only a small proportion of patients (5-19%) will respond to antihormonal therapy. ER-expression in ER-positive breast cancer can be assessed by positron emission tomography (PET) with [18F]fluoroestradiol (FES). In this study the investigators will evaluate whether FES-PET can be used to visualize and quantify ER-expression in ovarian cancer. If these results are positive, this would warrant further exploration of FES-PET imaging in ovarian cancer.

DETAILED DESCRIPTION:
Investigators will evaluate whether FES-PET can be used to visualize and quantify ER-expression in ovarian cancer. If these results are positive, this would warrant further exploration of FES-PET imaging in ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histological evidence or high clinical suspicion of epithelial ovarian cancer
2. The presence of at least one measurable lesion (RECIST version 1.1).
3. Histology or cytology can be obtained (may be ascites)
4. Eastern Cooperative Oncology Group performance status 0-2.
5. Postmenopausal status (defined as either >45 years with amenorrhea >12 months, or prior bilateral ovariectomy)
6. No history of other ER-positive malignancies
7. Signed written informed consent
8. Able to comply with the protocol

Exclusion Criteria:

1. Use of estrogen receptor ligands, including tamoxifen, fulvestrant or estrogens, during the 5 weeks before entry into the study
2. Life-expectancy ≤ 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The feasibility of FES-PET to visualize and quantify ER-positive lesions in epithelial ovarian cancer. | approximately 1 month
  Ovarian cancer patients planned for surgery or in which histology/cytology will be obtained, will undergo FES-PET/CT. FES-PET/CT will be qualitatively analyzed to determine whether ovarian cancer lesions can be visualized. FES-uptake will be quantified for all known lesions. Patient material will be stained for ER-expression to determine whether ER-positive metastases show FES-uptake.

SECONDARY OUTCOMES:
Correlation between FES-PET and immunohistochemistry (IHC) | approximately 1 month
  FES-uptake will be calculated for each lesions. Quantitative FES-uptake will be correlated to semi-quantitative IHC-scoring for ER-alpha, ER-bèta, and progesterone receptor.
Concordance between CT-scan and FES-PET | approximately 1 month
  CT-scan will be analyzed by a radiologist and lesions will classified into benign, equivocal and malignant lesions. FES-PET will be analyzed by a nuclear medicine physician and lesions will be classified. Concordance between FES-PET and CT-scan will be described. For discordant lesions, histology will be used as golden standard whenever available.

CONTACTS AND LOCATIONS:
Overall Officials: Geke AP Hospers, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Yoshida Y, Kurokawa T, Tsujikawa T, Okazawa H, Kotsuji F. Positron emission tomography in ovarian cancer: 18F-deoxy-glucose and 16alpha-18F-fluoro-17beta-estradiol PET. J Ovarian Res. 2009 Jun 16;2(1):7. doi: 10.1186/1757-2215-2-7. PMID 19527525
- [Background] Peterson LM, Mankoff DA, Lawton T, Yagle K, Schubert EK, Stekhova S, Gown A, Link JM, Tewson T, Krohn KA. Quantitative imaging of estrogen receptor expression in breast cancer with PET and 18F-fluoroestradiol. J Nucl Med. 2008 Mar;49(3):367-74. doi: 10.2967/jnumed.107.047506. Epub 2008 Feb 20. PMID 18287268